CLINICAL TRIAL: NCT04078503
Title: Neuroinflammation During ICU-associated Delirium in Critically Ill Patients and Its Association With Structural and Functional Brain Alterations: a Nested Case-control Study
Acronym: Delirium-fMRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: University of Pisa (Other); University of Turin, Italy (Other); University of Milano Bicocca (Other); Università degli Studi di Brescia (Other); Mie University (Other); Erasme University Hospital (Other); Maastricht University (Other)
Responsible Party: Principal Investigator, Piva Simone, Assistant Professor, Università degli Studi di Brescia
Other Study IDs: NP3468
Record Dates: First submitted 2019-03-30; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Delirium; Critical Illness
Keywords: neuroinflammation; fMRI; Functional MRI; ICU related delirium
MeSH Terms: conditions — Delirium; Critical Illness; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: All patients aspected to stay in ICU for at least 3 days who will develop delirium
- Control: All patients aspected to stay in ICU for at least 3 days who will not develop delirium (1:1 matched with the controls with a propensity score method).

SUMMARY:
With the present study, the authors aim to improve the knowledge of the pathophysiology of ICU-related delirium. In particular, the authors would like to clarify the possible correlation between neuroinflammation, evaluated longitudinally by serum dosage of 20 different neuroinflammation biomarkers, and brain structural and functional alterations (using brain fMRI).

DETAILED DESCRIPTION:
Pathophysiology of delirium is poorly understood; neuroinflammation and brain network disruption are claimed as possible causes of delirium.

The authors want to clarify the role of the alterations of different cellular components of neuroinflammation (neurons, glial cells, and endothelium) in delirium development. Moreover, the authors want to understand whether the neuroinflammation process could cause permanent structural and functional brain damage.

In a nested cross-sectional longitudinal case-control observational study in ICU admitted patients.

The objectives of the studies are as follow: 1) Neuroinflammation biomarkers evaluation in non-neurological ICU patients who develop delirium during ICU-stay (case) compared to matched non-delirious ICU patients (control), and 2) their correlation with brain structural and functional alterations evaluated with a resting-state fMRI protocol and PET.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* All patients admitted that would be expected to stay in ICU for at least 3 days

Exclusion Criteria:

* Acute neurological condition
* Chronic neurological condition (i.e., seizures, stroke, muscular illness).
* Hematological malignancy or immunological disease.
* Blood transfusion in the last 2 weeks
* Ongoing sedation
* Any condition which contraindicates MRI execution (presence of non-compatible devices or hemodynamic or respiratory instability).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll 30 critically ill patients in the study (case) matched to 30 controls (see sample size calculation).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2021-03-25 (Estimated); Study Completion 2021-06-25 (Estimated)

PRIMARY OUTCOMES:
Serum Neuroinflammation biomarkers in patients developing delirium. | 15 days
  Comparison of neuroinflammation biomarkers in patients developing delirium vs patients who do not develop delirium.

SECONDARY OUTCOMES:
fMRI alteration | 6 months
  Evaluation of brain functional alterations during delirium development (evaluated through resting state fMRI).
Correlation between biomarkers alterations and fMRI alterations | 15 days
  Evaluation of the correlation between serum neuroinflammation biomarkers alteration during delirium development and the alterations noted in during resting state fMRI

CONTACTS AND LOCATIONS:
Locations (1):
- Spedali Civili di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Yes
The database is in RedCap. We could share all data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Already available